CLINICAL TRIAL: NCT04647214
Title: ARGOS - A Phase IV, Prospective, 18-month Study to Assess the Effectiveness and Safety of Bimatoprost Intracameral Implant (DURYSTA) in US Clinical Practice
Brief Title: 18 Month Prospective Efficacy and Safety Study of Bimatoprost Intracameral Implant (DURYSTA)
Acronym: ARGOS
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MED-MA-EYE-0648
Record Dates: First submitted 2020-11-23; First posted 2020-11-30 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bimatoprost intracameral implant (DURYSTA) 10μg: Patients with OAG or OHT who are scheduled for intracameral administration of a bimatoprost intracameral implant by their ophthalmologist.

SUMMARY:
Study to collect effectiveness and safety data after administration of a bimatoprost intracameral implant in patients with open-angle glaucoma (OAG) or ocular hypertension (OHT).

ELIGIBILITY:
Inclusion Criteria:

- Patient diagnosed with OAG or OHT who is scheduled to receive a bimatoprost intracameral implant in at least one eye.

Exclusion Criteria:

- A history of any of the following ocular surgeries in the eye due to receive a bimatoprost intracameral implant:Ahmed Glaucoma Valve, Baerveldt shunt, Ex-Press glaucoma shunt implantation, Molteno shunt, Trabeculectomy, Vitrectomy, retinal surgery, CyPass Micro-Stent or Anterior Chamber Intraocular Lens (AC IOL) placement.

* Concurrent or anticipated enrollment in an interventional clinical trial involving either an investigational medicinal product or medical device.
* Previous enrollment in another Allergan bimatoprost intracameral implant study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include US patients with OAG or OHT who are scheduled for administration of a bimatoprost intracameral implant by their ophthalmologist.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of treated eyes that did not receive additional Intraocular Pressure (IOP) -lowering intervention/therapy per standard medical care | Baseline to Month 6
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.

SECONDARY OUTCOMES:
Proportion of treated eyes not receiving additional IOP-lowering intervention/therapy per standard medical care | Baseline to Month 4
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes not receiving additional IOP-lowering intervention/therapy per standard medical care | Baseline to Month 9
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes not receiving additional IOP-lowering intervention/therapy per standard medical care | Baseline to Month 12
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes not receiving additional IOP-lowering intervention/therapy per standard medical care | Baseline to Month 18
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Time from bimatoprost intracameral implant to first additional IOP-lowering intervention/therapy | Baseline to Month 18
  Time to first IOP-lowering intervention is defined as the time between treatment and IOP-lowering intervention.
Proportion of treated eyes achieving the predefined IOP outcomes without receiving additional IOP-lowering intervention/therapy | Baseline to Month 4
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes achieving the predefined IOP outcomes without receiving additional IOP-lowering intervention/therapy | Baseline to Month 6
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes achieving the predefined IOP outcomes without receiving additional IOP-lowering intervention/therapy | Baseline to Month 9
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes achieving the predefined IOP outcomes without receiving additional IOP-lowering intervention/therapy | Baseline to Month 12
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Proportion of treated eyes achieving predefined IOP outcomes without receiving additional IOP-lowering intervention/therapy | Baseline to Month 18
  IOP is a measurement of the fluid pressure inside the study eye. A negative change from baseline indicates an improvement and a positive change from baseline indicates a worsening.
Mean reduction in the number of topical IOP-lowering medications | Baseline to Month 4
  A numerical count by class of drug of topical IOP lowering medications being taken.
Mean reduction in the number of topical IOP-lowering medications | Baseline to Month 6
  A numerical count by class of drug of topical IOP lowering medications being taken.
Mean reduction in the number of topical IOP-lowering medications | Baseline to Month 9
  A numerical count by class of drug of topical IOP lowering medications being taken.
Mean reduction in the number of topical IOP-lowering medications | Baseline to Month 12
  A numerical count by class of drug of topical IOP lowering medications being taken.
Mean reduction in the number of topical IOP-lowering medications | Baseline to Month 18
  A numerical count by class of drug of topical IOP lowering medications being taken.
Proportion of treated eyes achieving complete success | Baseline to Month 4
  Complete success is defined as treated eyes with IOP <=18 mm Hg without any additional IOP lowering interventions/therapies after administration of the bimatoprost intracameral implant.
Proportion of treated eyes achieving complete success | Baseline to Month 6
  Complete success is defined as treated eyes with IOP <=18 mm Hg without any additional IOP lowering interventions/therapies after administration of the bimatoprost intracameral implant.
Proportion of treated eyes achieving complete success | Baseline to Month 9
  Complete success is defined as treated eyes with IOP <=18 mm Hg without any additional IOP lowering interventions/therapies after administration of the bimatoprost intracameral implant.
Proportion of treated eyes achieving complete success | Baseline to Month 12
  Complete success is defined as treated eyes with IOP <=18 mm Hg without any additional IOP lowering interventions/therapies after administration of the bimatoprost intracameral implant.
Proportion of treated eyes achieving complete success | Baseline to Month 18
  Complete success is defined as treated eyes with IOP <=18 mm Hg without any additional IOP lowering interventions/therapies after administration of the bimatoprost intracameral implant.
Proportion of treated eyes achieving qualified success | Baseline to Month 4
  Partial success is defined as treated eyes with IOP <=18 mm Hg with no Secondary Surgical Intervention (SSI) for glaucoma, while staying on the same or fewer topical IOP-lowering medications than baseline and or Selective Laser Trabeculoplasty (SLT), Argon Laser Trabeculoplasty (ALT) or MicroPulse Laser Trabeculoplasty (MLT).
Proportion of treated eyes achieving qualified success | Baseline to Month 6
  Partial success is defined as treated eyes with IOP <=18 mm Hg with no Secondary Surgical Intervention (SSI) for glaucoma, while staying on the same or fewer topical IOP-lowering medications than baseline and or Selective Laser Trabeculoplasty (SLT), Argon Laser Trabeculoplasty (ALT) or MicroPulse Laser Trabeculoplasty (MLT).
Proportion of treated eyes achieving qualified success | Baseline to Month 9
  Partial success is defined as treated eyes with IOP <=18 mm Hg with no Secondary Surgical Intervention (SSI) for glaucoma, while staying on the same or fewer topical IOP-lowering medications than baseline and or Selective Laser Trabeculoplasty (SLT), Argon Laser Trabeculoplasty (ALT) or MicroPulse Laser Trabeculoplasty (MLT).
Proportion of treated eyes achieving qualified success | Baseline to Month 12
  Partial success is defined as treated eyes with IOP <=18 mm Hg with no Secondary Surgical Intervention (SSI) for glaucoma, while staying on the same or fewer topical IOP-lowering medications than baseline and or Selective Laser Trabeculoplasty (SLT), Argon Laser Trabeculoplasty (ALT) or MicroPulse Laser Trabeculoplasty (MLT).
Proportion of treated eyes achieving qualified success | Baseline to Month 18
  Partial success is defined as treated eyes with IOP ≤18 mm Hg with no Secondary Surgical Intervention (SSI) for glaucoma, while staying on the same or fewer topical IOP-lowering medications than baseline and or Selective Laser Trabeculoplasty (SLT), Argon Laser Trabeculoplasty (ALT) or MicroPulse Laser Trabeculoplasty (MLT).
Number of participants experiencing treatment emergent adverse events | Baseline to Month 18

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (39):
- United States (39):
  - Angeles Eye Institute /ID# 240368, Culver City, California
  - Hamilton Glaucoma Center Shiley Eye Center UCSD /ID# 240364, La Jolla, California
  - American Institute of Research /ID# 247820, Los Angeles, California
  - North Bay Eye Associates Inc. /ID# 240362, Petaluma, California
  - Pacific Eye Associates /ID# 240536, San Francisco, California
  - Colorado Eye Institute /ID# 240798, Colorado Springs, Colorado
  - ICON Eye Care /ID# 240681, Grand Junction, Colorado
  - Eye Associates of Fort Meyers /ID# 244476, Fort Myers, Florida
  - MedEye Associates /ID# 240374, Miami, Florida
  - Center for Sight - Sarasota /ID# 244578, Sarasota, Florida
  - Newsom Eye & Laser Center /ID# 253287, Sebring, Florida
  - Dr. Andrew Gardner Logan, FL /ID# 240361, Tamarac, Florida
  - Your Eye Specialists /ID# 253286, Weston, Florida
  - Georgia Eye Partners /ID# 240061, Atlanta, Georgia
  - Kovach Eye Institute /ID# 244581, Elmhurst, Illinois
  - Stiles Eyecare Excellence /ID# 240376, Overland Park, Kansas
  - The Eye Care Institute /ID# 240367, Louisville, Kentucky
  - John Hopkins Wilmer Eye Institute /ID# 243701, Bethesda, Maryland
  - Midwest Vision Research Foundation at Pepose Vision Institute /ID# 240537, Chesterfield, Missouri
  - Wiles Eye Center /ID# 240808, Kansas City, Missouri
  - Ophthalmology Associates /ID# 240799, St Louis, Missouri
  - Eye Associates of North Jersey /ID# 244585, Dover, New Jersey
  - Hudson Eye /ID# 240805, Jersey City, New Jersey
  - Glaucoma Care Center /ID# 252021, Livingston, New Jersey
  - Burlington County Eye Physicians /ID# 244594, Willingboro, New Jersey
  - MaculaCare PLLC /ID# 244593, New York, New York
  - New York New Jersey Eye Institute /ID# 244590, Orangeburg, New York
  - New York Eye Surgery Associates, PLLC /ID# 244592, The Bronx, New York
  - Duke Eye Center /ID# 244478, Durham, North Carolina
  - Bergstrom Eye Research LLC /ID# 240363, Fargo, North Dakota
  - META Medical Research Institute, LLC /ID# 240800, Dayton, Ohio
  - Oklahoma Eye Surgeons /ID# 240373, Oklahoma City, Oklahoma
  - Scott and Christie and Associates /ID# 244574, Cranberry Township, Pennsylvania
  - Vanderbilt University Medical Center /ID# 244577, Nashville, Tennessee
  - Glaucoma Associates of Texas /ID# 240682, Dallas, Texas
  - Glaucoma Associates of Texas /ID# 253289, Dallas, Texas
  - El Paso Eye Surgeons, P.A. /ID# 240366, El Paso, Texas
  - DCT Shah Eye Research Institut /ID# 240375, Mission, Texas
  - The Eye Centers of Racine and Kenosha LTD /ID# 240059, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mann E, Kammer JA, Sawhney G, An J, Werts EC, Vera V, Rivas M, Lai H, Sonparote S, Craven ER. Prospective 18-Month Study of Bimatoprost Intracameral Implant in Patients with Open-Angle Glaucoma or Ocular Hypertension in US Clinical Practice. Drugs. 2025 Mar;85(3):397-414. doi: 10.1007/s40265-025-02157-1. Epub 2025 Feb 13. PMID 39946034
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=MED-MA-EYE-0648#additional-resources-section